CLINICAL TRIAL: NCT00171925
Title: Therapy With Zoledronic Acid in Patients With Multiple Myeloma Stage I
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment in study could not be reached after 8 yrs of recruiting
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446 DE01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Myeloma Stage I
Keywords: Multiple Myeloma; Stage I; Zoledronic acid; Progression
MeSH Terms: conditions — Multiple Myeloma; Disease Progression | interventions — Zoledronic Acid; Calcium; Vitamin D

ARMS (2):
- Zoledronic acid (ZOL446) (Experimental): Participants received intravenous infusion of Zoledronic acid every 4 weeks for 48 weeks, and calcium and Vitamin D daily.
  Interventions: Drug: Zoledronic acid; Dietary Supplement: Calcium / Vitamin D
- Control (No Intervention): No treatment with study medication.

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid administered via normal saline intravenous infusion (over 15 minutes) every 4 weeks. Dosage was according to calculated creatinine clearance: patients with baseline creatinine clearance > 60 ml/min received 4 mg; for patients with mild to moderate renal impairment, doses were calculated to achieve the same AUC as that achieved in patients with creatinine clearance of 75 ml/min, assuming target AUC of 0.66 (mg*hr/l).
  Arms: Zoledronic acid (ZOL446)
Dietary Supplement: Calcium / Vitamin D — Patients on zoledronic acid received 500 mg calcium and 400-500 IU vitamin D combination tablet daily.
  Arms: Zoledronic acid (ZOL446)

SUMMARY:
Multiple myeloma is a disease of B-lymphocytes producing malignant plasma cells. Malignant plasma cells induce osteolytic lesions, which is characteristic for progression of multiple myeloma. It is the aim of this study to investigate whether zoledronic acid has an influence on the progression of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria

* Evidence of myeloma according to the criteria of the British Columbia Cancer Agency (for the diagnosis, 2 of the 3 criteria must be met):

  * Evidence of paraprotein in the serum or urine
  * Bone marrow infiltration with plasma cells which represent more than 10% of the nucleated cells
  * Radiologically, at least one osteolytic lesion
* Asymptomatic patients with Stage I (Durie and Salmon) multiple myeloma

Exclusion criteria:

* Patients with more than one osteolytic lesion on conventional skeletal radiography
* Previous treatment with bisphosphonates
* bilirubin > 2.5 mg/dl
* Abnormal renal function as evidenced by: A calculated creatinine clearance < 30 ml/minute. Creatinine clearance (CrCl) is calculated using the Cockcroft-Gault formula:

  * CrCl= [140-age(years)] x weight(kg)/[72xserumcreatinine(mg/dL)] X {0.85 for female patients}
* Patients with other malignant diseases or severe concomitant diseases
* Potentially fertile patients who are not using a reliable and appropriate method of contraception
* Pregnancy or breast-feeding
* Participation in another clinical study with an investigational drug within 12 weeks of study entry
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants)

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2000-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid (ZOL446) | Control
Started | 72 | 71
Completed | 42 | 40
Not Completed | 30 | 31
Not completed — Adverse Event | 10 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Administrative problems | 10 | 11
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid (ZOL446) | Control | Total
Number analyzed (Participants) | 72 | 71 | 143
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (12.02) | 62.1 (10.79) | 60.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 31 | 73
  Male | 30 | 40 | 70
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 69 | 70 | 139
  Oriental | 2 | 0 | 2
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Germany | 72 | 71 | 143

OUTCOME MEASURES:

1. Primary Outcome: Days of Progression Free Survival
Description: Progression-free survival was defined as time from date of randomization to death from any cause or one of the following events:
  * progression to stage II or III according to Salmon & Durie classification
  * skeletal related events (pathologic fracture, initiation of radiotherapy or surgery on bone, spinal cord compression or hypercalcemia)
  * unequivocal progression of osteolytic lesions (at least a 20% increase in the largest diameter of one existing osteolytic lesion which is measured in at least one dimension as 20 mm with conventional techniques), determined radiologically.
Time Frame: 48 months
Population: Intent to Treat Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Zoledronic Acid (ZOL446) | Control
Number analyzed (Participants) | 71 | 69
Days | 1078.1 (59.53) | 992.80 (61.83)

2. Secondary Outcome: Number of Patients With Progression by Individual Criteria
Description: Number of patients with progression by individual criteria consisting of Progression of disease overall, Skeletal-related events (including pathological fracture, initiation of radiotherapy or surgery on bone, spinal cord compression or Hypercalcemia), Progression to stage II or III according to Salmon & Durie classification, and unequivocal progression of osteolytic lesion. Patients are counted separately for every type of progression, but only once for Overall Progression.
Time Frame: 48 months
Population: Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid (ZOL446) | Control
Number analyzed (Participants) | 71 | 69
Participants
  Progression of disease overall | 19 | 26
  Skeletal-related events | 0 | 4
  Progression to stage II or III | 17 | 24
  Unequivocal progression of osteolytic lesion | 3 | 10

3. Secondary Outcome: The Number of Participants With the Development of Skeletal Complications
Description: * Pathologic fracture: bone fractures that occur spontaneously or from trivial trauma. New vertebral compression fracture defined as a decrease in vertebral height of 25% from baseline
  * Spinal cord compression: the impingement of tumor on the spinal cord confirmed by radiography
  * Bone Radiotherapy: Bone irradiation to palliate painful lesions, treat or prevent pathologic fractures or spinal cord compression
  * Surgery on bone: surgical procedures performed to set, stabilize or prevent pathologic fractures or areas of spinal cord compression
  * Hypercalcemia: Corrected serum calcium ≥ 12.0 mg/dl
Time Frame: 48 months
Population: Intent to treat population
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid (ZOL446) | Control
Number analyzed (Participants) | 71 | 69
Participants
  Skeletal events overall | 0 | 4
  Pathological fracture | 0 | 1
  Initiation of radiotherapy or surgery on bone | 0 | 1
  Spinal cord compression | 0 | 2
  Hypercalcemia | 0 | 0

ADVERSE EVENTS:
Groups:
- Zoledronic Acid: Participants received intravenous infusion of Zoledronic acid every 4 weeks for 48 weeks, and calcium and Vitamin D daily.
Arm/Group | Zoledronic Acid | Control
Serious Adverse Events (participants affected / at risk) | 28/72 | 12/71
Other Adverse Events (participants affected / at risk) | 61/72 | 51/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=72) | Control (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac amyloidosis (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteonecrosis of the jaw (Musculoskeletal and connective tissue disorders) | 4 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 2 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Stupor (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Uterine malposition (Reproductive system and breast disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=72) | Control (N=71)
Vertigo (Ear and labyrinth disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Nausea (Gastrointestinal disorders) | 6 | 2
Chills (General disorders) | 5 | 0
Fatigue (General disorders) | 7 | 3
Influenza like illness (General disorders) | 7 | 0
Oedema peripheral (General disorders) | 4 | 3
Pain (General disorders) | 5 | 4
Pyrexia (General disorders) | 11 | 0
Bronchitis (Infections and infestations) | 7 | 4
Infection (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 24 | 10
Respiratory tract infection (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 4 | 1
Blood creatinine increased (Investigations) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7
Headache (Nervous system disorders) | 11 | 5
Depression (Psychiatric disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 2
Hypertension (Vascular disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
Only exploratory analyses were performed as the trial was terminated early due to lack of obtaining the required sample size. Secondary Outcomes for Quality of Life and Bone Markers not posted due to sparse data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.